CLINICAL TRIAL: NCT01998945
Title: Back on My Feet: Emotional Recovery From Fall Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nimali Jayasinghe, Assistant Professor of Psychology, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1306014003; K23MH090244 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-12-03 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Posttraumatic Stress Disorder; Subsyndromal Posttraumatic Stress Disorder; Fear of Falling
Keywords: Exposure therapy; Cognitive behavioral therapy; Relaxation Training; Older Adults; Fall Injury; Anxiety; Posttraumatic Stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exposure-based Cognitive Behavioral Therapy (ET) (Experimental): Participants will receive exposure-based cognitive behavioral therapy
  Interventions: Behavioral: Exposure-based Cognitive Behavioral Therapy
- Relaxation Training (RT) (Active Comparator): Participants will receive relaxation training
  Interventions: Behavioral: Relaxation Training

INTERVENTIONS:
Behavioral: Exposure-based Cognitive Behavioral Therapy — Eight 75-minute, in-home sessions delivered twice weekly for 4 weeks of exposure-based cognitive behavioral therapy, a time-limited treatment that focuses on confronting avoided memories and situations and identifying and managing distressing thoughts.
  Arms: Exposure-based Cognitive Behavioral Therapy (ET)
Behavioral: Relaxation Training — Eight 75-minute, in-home sessions delivered twice weekly for 4 weeks of Relaxation Training, that focus on muscle relaxation and diaphragmatic breathing to address the physical symptoms of anxiety.
  Arms: Relaxation Training (RT)

SUMMARY:
We will compare two programs that are designed to help older adults who have had fall injuries manage anxiety and improve their level of functioning. We expect that both programs will provide some benefit, but that one will promote better management.

DETAILED DESCRIPTION:
Fall accidents can be frightening experiences that cause life-changing injuries. Each year, millions of older Americans who fall may develop disabling anxiety and related distress, functional limitations, and poor health.

Our previous study adapted a well-researched anxiety treatment, Exposure-based Cognitive Behavioral Therapy (ET), for older adults diagnosed with full posttraumatic stress disorder (PTSD), subsyndromal PTSD, or fear of falling after fall injury. The approach was well-accepted by subjects and they reported both reductions in anxiety and having more fully returned to normal living immediately after the treatment and then three months later.

The purpose of this pilot study is to compare ET to another active treatment, Relaxation Training (RT). Both study treatments will consist of eight home-based sessions. ET consists of education about anxiety, relaxation training, managing distressing thoughts, healthy routine, and confronting avoided memories and situations. RT consists of techniques to ease bodily tension.

Twenty-four subjects will be randomly assigned to one of the two treatment groups. The study will compare how subjects in each group improve on outcomes such as diagnosis, anxiety severity, and quality of life over the course of treatment, and at three- and six-month follow-up.

The findings will provide the basis for larger future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older
* Fall accident requiring emergency room or inpatient hospital medical care with return home within past nine months
* Community dwelling
* Able to ambulate independently or with an assistive device
* English-speaking
* Diagnosis of PTSD, subsyndromal PTSD, or Fear of Falling (determined by interview)

Exclusion Criteria:

* Cognitive impairment
* Serious or terminal illness
* Aphasia
* Current substance abuse
* Lifetime history of psychotic disorder and/or bipolar disorder
* Active suicidal or homicidal ideation
* Prescription psychotropic medication begun < 6 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline clinician-rated PTSD at 6 weeks | Baseline, Week 6

SECONDARY OUTCOMES:
Change from baseline fear of falling at 6 weeks | Baseline, Week 6
Change from baseline depression at 6 weeks | Baseline, Week 6
Change from baseline anxiety at 6 weeks | Baseline, Week 6
Change from baseline self-reported PTSD at 6 weeks | Baseline, Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Nimali Jayasinghe, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States